CLINICAL TRIAL: NCT06994260
Title: Multispectral Optoacoustic Tomography (MSOT) and Ultrasound Localization Microscopy (ULM) as Diagnostic Imaging for Lymphatic, Venous and Arteriovenous Malformations
Brief Title: Diagnostic Imaging of Vascular Malformations Using MSOT and ULM
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Erlangen (Other)
Collaborators: PD Dr. med. Ferdinand Knieling, Department of pediatrics, University of Erlangen-Nürnberg (Unknown)
Responsible Party: Principal Investigator, Ulrich Rother, Senior Consultant, Department of Vascular Surgery, University Hospital Erlangen, University Hospital Erlangen
Other Study IDs: MSOT_ULM_malfo
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Vascular Malformation; Arteriovenous Malformation; Lymphatic Malformation; Venous Malformations
Keywords: Vascular Malformation; Venous Malformation; Arteriovenous Malformation; Lymphatic Malformation; MSOT; ULM
MeSH Terms: conditions — Vascular Malformations; Arteriovenous Malformations; Lymphatic Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Venous Malformation: Patients with venous malformations.
  Interventions: Diagnostic Test: Multispectral Optoacoustic Tomography; Diagnostic Test: Ultrasound Localization Microscopy
- Arteriovenous Malformations: Patients with arteriovenous malformations.
  Interventions: Diagnostic Test: Multispectral Optoacoustic Tomography; Diagnostic Test: Ultrasound Localization Microscopy
- Lymphatic Malformations: Patients with lymphatic malformations.
  Interventions: Diagnostic Test: Multispectral Optoacoustic Tomography; Diagnostic Test: Ultrasound Localization Microscopy

INTERVENTIONS:
Diagnostic Test: Multispectral Optoacoustic Tomography — MSOT is an advanced imaging technology that combines laser-induced ultrasound and light absorption to visualize biological tissues. By detecting ultrasound waves generated from tissue absorption of multispectral light, MSOT provides high-resolution, real-time images with functional and molecular information. One of its use is in biomedical research and clinical applications to study blood oxygenation and tissue composition, making it valuable for areas such as vascular research.
  In this study, we aim to utilize MSOT to differentiate between venous, arteriovenous and lymphatic malformations.
Diagnostic Test: Ultrasound Localization Microscopy — ULM is a cutting-edge imaging technique that significantly enhances the resolution of traditional ultrasound by tracking the movement of microbubble contrast agents within blood vessels. This approach enables the visualization of microvascular structures and blood flow dynamics at a super-resolution scale, beyond the diffraction limit of conventional ultrasound.
  In this study, we aim to utilize ULM to differentiate between venous, arteriovenous and lymphatic malformations.

SUMMARY:
This clinical study evaluates the efficacy and accuracy of Multispectral Optoacoustic Tomography (MSOT) and Ultrasound Localization Microscopy (ULM) for imaging and diagnosing vascular malformations (venous, arteriovenous, lymphatic). The study aims to enhance diagnostic precision and improve treatment planning through advanced non-invasive imaging techniques.

DETAILED DESCRIPTION:
This study aims to investigate whether Multispectral Optoacoustic Tomography (MSOT) and Ultrasound Localization Microscopy (ULM) can accurately differentiate between lymphatic, venous, and arteriovenous vascular malformations. MSOT can determine oxygen levels based on the expected low oxygen content in venous blood, high oxygen content in arterial blood, and the absence of oxygen in lymphatic fluid. Additionally, ULM, utilizing microbubbles, measures blood flow velocities, which may help identify and distinguish these malformations or their mixed forms.

To date, vascular malformations of blood and lymphatic vessels are commonly diagnosed using cross-sectional imaging techniques such as ultrasound, computed tomography (CT), or magnetic resonance imaging (MRI). MSOT introduces a novel, non-invasive diagnostic approach that enables the assessment of oxygenated hemoglobin concentrations and oxygen levels in blood and tissue. Previous studies (e.g., MSOT_IC, MSOT_PI) demonstrated the capability of MSOT to visualize muscle perfusion in patients with peripheral arterial disease. Moreover, it has successfully identified muscle structures and the clinical severity of Duchenne muscular dystrophy by detecting endogenous biomarkers like collagen and lipids.

The objective of this study is to utilize MSOT and ULM as supplementary diagnostic tools to conventional imaging methods to accurately identify and distinguish between venous, arteriovenous, and lymphatic malformations in patients. This approach has the potential to reduce exposure to ionizing radiation from CT scans and minimize the need for resource-intensive MRI procedures in the future.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed vascular malformations (arteriovenous, venous, or lymphatic).
* ≥18 years old and able to give their consent

Exclusion Criteria:

* No imaging for diagnostic confirmation has been performed or is planned.
* Lack of written consent
* <18 years old
* Safety concerns of the study physician (a patient with physical, psychological, or psychiatric conditions that, in the opinion of the study physician, could compromise the patient's safety or the quality of the data, thereby making the patient an unsuitable candidate for the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients (≥18 years old) with diagnosed vascular malformations. These may be of lymphatic, venous, or arteriovenous origin.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative signal of total hemoglobin (HbT), oxygenated hemoglobin (HbO2), deoxygenated hemoglobin (Hb), and oxygen saturation (mSO2). | through study completion, an average of 1 year
  using MSOT
Quantification of perfusion dynamics in the respective vessel. | through study completion, an average of 1 year
  using ULM

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Erlangen, Department of Vascular Surgery, Erlangen, Bavaria, Germany

REFERENCES:
- [Background] Seront E, Vikkula M, Boon LM. Venous Malformations of the Head and Neck. Otolaryngol Clin North Am. 2018 Feb;51(1):173-184. doi: 10.1016/j.otc.2017.09.003. PMID 29217061
- [Background] Kansy K, Bodem J, Engel M, Freudlsperger C, Mohlenbruch MA, Herweh C, Bendszus M, Hoffmann J, Kargus S. Interdisciplinary treatment algorithm for facial high-flow arteriovenous malformations, and review of the literature. J Craniomaxillofac Surg. 2018 May;46(5):765-772. doi: 10.1016/j.jcms.2018.03.002. Epub 2018 Mar 9. PMID 29609843
- [Background] Gray RL, Ortiz RA, Bastidas N. Combined Surgery and Intraoperative Sclerotherapy for Vascular Malformations of the Head/Neck: The Hybrid Approach. Ann Plast Surg. 2018 Apr;80(4 Suppl 4):S156-S157. doi: 10.1097/SAP.0000000000001366. PMID 29596084
- [Background] Dompmartin A, Vikkula M, Boon LM. Venous malformation: update on aetiopathogenesis, diagnosis and management. Phlebology. 2010 Oct;25(5):224-35. doi: 10.1258/phleb.2009.009041. PMID 20870869
- [Background] Demene C, Robin J, Dizeux A, Heiles B, Pernot M, Tanter M, Perren F. Transcranial ultrafast ultrasound localization microscopy of brain vasculature in patients. Nat Biomed Eng. 2021 Mar;5(3):219-228. doi: 10.1038/s41551-021-00697-x. Epub 2021 Mar 15. PMID 33723412
- [Background] Carqueja IM, Sousa J, Mansilha A. Vascular malformations: classification, diagnosis and treatment. Int Angiol. 2018 Apr;37(2):127-142. doi: 10.23736/S0392-9590.18.03961-5. Epub 2018 Feb 8. PMID 29424187